CLINICAL TRIAL: NCT00858338
Title: Phase-II Study of Adjuvant Intraperitoneal FUDR Treatment Added to Chemoradiation (5-fluorouracil/Leucovorin Plus Total Dose 4500 cGy of External Beam Radiotherapy) in Patients With Fully Resected Locally Advanced Gastric Adenocarcinoma (R0 Resection and at Least D1 Lymph-node Dissection)
Brief Title: Adjuvant Intraperitoneal Floxuridine Added to Chemoradiation for Fully Resected Advanced Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Franco Muggia, MD, NYU Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-51 (H 10610); NCT00058916 (obsolete NCT alias)
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Gastric Cancer; Stomach Cancer
Keywords: stomach cancer; gastroesophageal junction cancer; GEJ cancer; intraperitoneal; adjuvant chemoradiation therapy; resection of advanced stomach cancer; locally advanced stomach cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Floxuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Potentially curative surgery — Surgery:
  Week 1: Potentially curative surgery. If the tumor successfully resected (microscopically disease-free margins, Ro, with regional lymphadenectomy for proper staging), the ip catheter in place.
  Weeks 2-4: Recovery. Then continue to adjuvant IP chemotherapy.
Drug: Floxuridine (IP) — Adjuvant IP Chemotherapy:
  week 1: ip Floxuridine 3 gm/day, days 1,2,3. week 2: 1 week without treatment. week 3: ip Floxuridine 3 gm/day protocol days 15,16,17. week 4: 1 week without treatment. Then continue to chemoradiation therapy.
  Other Names: FUDR
Procedure: Adjuvant Chemoradiation therapy — Adjuvant Chemoradiation therapy:
  week 1: 5-FU 425 mg/m2/day x 5 days + Leucovorin (LV) 20 mg/m2/day x 5days; weeks 2-4: recovery; weeks 5-9: radiation, 150 cGy x 5 fractions/week x 5 weeks; week 5: 5-FU 400 mg/m2 + LV 20 mg/m2 each day on days 1-4; week 9: 5-FU 400 mg/m2 + LV 20 mg/m2 each day on days 1-3; week 14: 5-FU 425 mg/m2/day x 5 days + Leucovorin (LV) 20 mg/m2/day x 5days; week 19: 5-FU 425 mg/m2/day x 5 days + Leucovorin (LV) 20 mg/m2/day x 5days.

SUMMARY:
This study is to evaluate the efficacy and safety of addition of intraperitoneal (ip) Floxuridine to adjuvant chemoradiation therapy for patients under-going potentially curative stomach resection.

DETAILED DESCRIPTION:
Most patients diagnosed with stomach cancer in the US fail to be cured by gastric resection, and most trials of adjuvant chemotherapy do not improve survival rates. However, it has shown that chemo-radiotherapy can substantially increase survival rates after gastric resection in a recent intergroup randomized study (INT 0116) that used adjuvant chemoradiation of 5-fluorouracil (5-FU) and leucovorin concurrently with total dose of 4500 cGy of external-beam radiation treatment (RT) to the abdominal tumor nodal field in patients with resected, locally advanced gastric cancer. However, since the most common recurrences in both arms (surgery only vs. surgery followed by chemoradiation) were regional, typically abdominal carcinomatosis, this may indicate the need for adjuvant ip floxuridine to be added to adjuvant chemoradiation. Our experience for ip floxuridine leads us to hypothesize that the addition of this type of therapy to adjuvant chemoradiation may further increase the cure-rate for patient under-going potentially curative gastric resection. It seems important to convincingly demonstrate the effect of ip floxuridine treatment combined with the chemoradiation regimen. This became the basis for the design of this Phase II study, which will test the toxicity and efficacy of ip floxuridine added to chemo-radiation of the INT 0116 study. The protocol is to be completed in three years, and it may become a springboard for planning and initiation of a pivotal multi-institutional trials.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility to the protocol is established following complete evaluation specified under 9.2 of the study protocol. This evaluation includes the diagnosis and disease stage. Untreated patients with histologically documented gastric/GEJ carcinoma stages IB-IV (Mo), become eligible.
* Patients who underwent emergency surgery for indications such as gastrointestinal obstruction, perforation or hemorrhage, or patients with surgery already performed, are eligible as long as the surgery is considered curative (Ro) as specified in section 9.3 of the study protocol.
* A device for adjuvant ip chemotherapy has to be in situ, placed during the surgery or early (1-3 weeks) thereafter. Time elapsed since the surgery must not exceed 4 weeks.
* Patient's diagnosis and staging, based on postoperative pathological findings, has to confirm stage IB-IV Mo adenocarcinoma of the stomach or GEJ. Patients and their clinical records must be evaluated by protocol surgical, radiation and medical oncologists, and sections of resected primary tumor and lymph nodes by protocol surgical pathologist.
* Each patient has to undergo pretreatment evaluation, sign Informed Consent, and be registered.
* Patients at least 18 years of age with performance status 0-2 (Appendix B of the study protocol).
* An adequate bone-marrow reserve (segmented neutrophils and bands, at least 1,500/ mmL, thrombocytes at least 100,000 /mmL, hemoglobin at least 9 gm/dL).
* Preserved liver and renal function (total serum bilirubin <2 mg/dL, SGOT/SGPT not greater than 2.5x the upper limit of normal, alkaline phosphatase not greater than 2.5x the upper limit of normal, BUN not greater than 30 mg/dL, creatinine concentration not greater than 1.5 mg/dL or creatinine clearance >60 mL/min), and negative BHcG in females of reproductive potential, are required.
* Patient must have evidence of at least unilateral renal function as established by CT scan with contrast or nephrogram. If only one kidney is present, at least two thirds of the functioning kidney must be excluded from any radiation port.
* The prothrombin time, activated partial thromboplastin time, and thrombin time should be within the range of normal values.
* All patients and records must be evaluated by a Surgical, Radiation and Medical Oncologists within one month before their entry to this protocol. There should be a reasonable assurance that patient will be available for planned post-treatment follow-up.
* Each patient must sign the Informed Consent Form.

Exclusion Criteria:

* Patients who do not meet criteria specified in inclusion criteria, and patients who have received prior RT, chemotherapy or immunotherapy.
* Patients with another active invasive malignancy. Adequately treated basal cell or squamous cell skin cancer, in-situ cervix cancer, or other cancers the patient has been free for at least 5 years, are acceptable.
* Patients with active or uncontrolled infection including HIV.
* Patients with psychiatric disorders that would interfere with their consent.
* Pregnant and nursing patients. Patients of reproductive age may not participate unless they agree to use an effective contraceptive method.
* Patients with any other severe concurrent disease, which in judgment of protocol investigators would make the patient inappropriate for this study.
* Protocol patients who did not receive ip FUDR treatment for complications related to catheter insertion or maintenance. However, these patients may still undergo off-protocol chemoradiation.
* Patients who did not sign written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-12; Primary Completion 2007-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
toxicity of IP FUDR after surgery prior to chemoradiation | 6 months

SECONDARY OUTCOMES:
overall survival | up to 10 years
  every 4 months the first year after treatment; every 6 months 2nd and 3rd year; yearly thereafter up to a total 10 years
Time to relapse, disease specific survival | up to 10 years
  every 4 months the first year after treatment; every 6 months 2nd and 3rd year; yearly thereafter up to a total 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Bellevue Hospital, New York, New York
  - NYU Cancer Center, New York, New York
  - NYU Tisch Hospital, New York, New York

REFERENCES:
- See also: Publication for this study — http://www.ncbi.nlm.nih.gov/pubmed/21769462